CLINICAL TRIAL: NCT00438490
Title: Phase 2 Study of Recombinant Human Prolactin Efficacy and Safety
Brief Title: The Safety and Efficacy of Recombinant Human Prolactin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Corrine Welt, Associate Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2001-P-001057
Record Dates: First submitted 2007-02-20; First posted 2007-02-22 (Estimated); Results first posted 2013-04-18 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2017-12

CONDITIONS: Healthy
Keywords: galactorrhea; prolactin; bone turnover; menstrual cycle; Control Groups; Women
MeSH Terms: conditions — Galactorrhea

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- recombinant human prolactin (Experimental): Recombinant Human Prolactin 60 mcg/kg once daily subcutaneous injection
  Interventions: Drug: Recombinant Human Prolactin
- Placebo (Placebo Comparator): Normal saline placebo subcutaneous injection
  Interventions: Drug: Recombinant Human Prolactin

INTERVENTIONS:
Drug: Recombinant Human Prolactin

SUMMARY:
Medications used to increase breast milk production increase prolactin secretion, the main hormone of lactation. There are no FDA approved medications used to improve breast feeding, but metoclopramide is used off-label and can have intolerable side effects. We examined the biological activity and safety of recombinant human prolactin (r-hPRL) as a potential medication to augment lactation. In this study, the effect of r-hPRL on breast milk production in women who did not recently deliver a baby and its effect on the bones and menstrual cycle were tested.

DETAILED DESCRIPTION:
There are no FDA approved medications in the U.S. to augment lactation. Metoclopramide is used off-label but can have intolerable side effects. We examined the biological activity and safety of recombinant human prolactin (r-hPRL) as preliminary data for its use to augment lactation. Healthy, non-postpartum women (n=21) with regular menstrual cycles underwent a 7 day randomized, double-blind, placebo-controlled trial of r-hPRL. Galactorrhea, markers of bone turnover, calcium homeostasis and gonadal function were measured and side effects recorded.

ELIGIBILITY:
Inclusion Criteria:

Healthy Subjects will meet the following criteria:

1. 18 to 40 years of age
2. Normal weight (BMI 17 to £ 30 kg/m2)
3. Good general health
4. On no medications for at least 3 months before the study
5. Regular menstrual cycles every 25-35 days with ovulation documented by a luteal phase progesterone level
6. No evidence of androgen excess
7. Normal TSH, prolactin and hematocrit
8. No current interest in conception
9. No history of osteoporosis
10. No use of medications known to affect bone turnover
11. No alcoholism
12. No smoking
13. No history of medical problems or treatment known to affect bone turnover.

Exclusion Criteria:

Subjects will be excluded for pregnancy or evidence of breast masses.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2002-04; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corrine K. Welt, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Corrine Welt, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Page-Wilson G, Smith PC, Welt CK. Short-term prolactin administration causes expressible galactorrhea but does not affect bone turnover: pilot data for a new lactation agent. Int Breastfeed J. 2007 Jul 24;2:10. doi: 10.1186/1746-4358-2-10. PMID 17650319

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Normal Saline Placebo once daily
- Recombinant Human Prolactin: Recombinant Human Prolactin 60 mcg/kg once daily
Period: Overall Study
Arm/Group | Placebo | Recombinant Human Prolactin
Started | 12 | 9
Completed | 12 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Recombinant Human Prolactin: RhProlactin once daily
  Recombinant Human Prolactin :
- Total: Total of all reporting groups
Arm/Group | Placebo | Recombinant Human Prolactin | Total
Number analyzed (Participants) | 12 | 9 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 9 | 21
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.1 (4.0) | 27.9 (6.4) | 28.4 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 9 | 21
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 9 | 21

OUTCOME MEASURES:

1. Primary Outcome: Galactorrhea
Description: Galactorrhea is breast milk production.
Time Frame: 7 days
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Recombinant Human Prolactin
Number analyzed (Participants) | 12 | 9
percentage of participants | 0 | 56

2. Secondary Outcome: N-telopeptide
Time Frame: 7 days
Measure: Mean (Standard Error); unit: nM/mM
Groups:
- Recombinant Human Prolactin: Recombinant Human Prolactin 60 mcg/kg once daily subcutaneous injection
  Recombinant Human Prolactin
- Placebo: Normal saline placebo subcutaneous injection
  Recombinant Human Prolactin
Arm/Group | Recombinant Human Prolactin | Placebo
Number analyzed (Participants) | 9 | 12
nM/mM | 7.4 (1.8) | 6.9 (0.7)

3. Secondary Outcome: Menstrual Cycle Length
Time Frame: 28 days
Measure: Mean (Standard Error); unit: Days
Arm/Group | Placebo | Recombinant Human Prolactin
Number analyzed (Participants) | 12 | 9
Days | 28.8 (1.0) | 30.1 (1.1)

4. Secondary Outcome: Estradiol
Time Frame: 7 days
Measure: Mean (Standard Error); unit: pmol/L
Arm/Group | Placebo | Recombinant Human Prolactin
Number analyzed (Participants) | 12 | 9
pmol/L | 634 (175) | 467 (72)

ADVERSE EVENTS:
Time Frame: Course of the entire study
Groups:
- Placebo: Placebo
Arm/Group | Placebo | Recombinant Human Prolactin
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/9
Other Adverse Events (participants affected / at risk) | 9/12 | 3/9
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=12) | Recombinant Human Prolactin (N=9)
fatigue (General disorders) | 1 (1) | 1 (1)
moodiness (General disorders) | 0 (0) | 1 (1)
Enlarged Lymph node (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Headache (General disorders) | 3 (3) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0)
Bruising from blood draw (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes